CLINICAL TRIAL: NCT06194344
Title: The Effectiveness of Individualized Imagery Scripts on Sleep, Psychosis, and Suicidality Among Inpatients With Psychosis: A Randomized Control Pilot Study
Brief Title: The Effectiveness of Individualized Imagery Scripts on Sleep, Psychosis, and Suicidality Among Inpatients With Psychosis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Alia Warner, Associate Warner, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HSC-MS-23-0915
Record Dates: First submitted 2023-12-08; First posted 2024-01-08 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Psychosis
Keywords: sleep therapy; suicidality; psychosis
MeSH Terms: conditions — Psychotic Disorders; Suicidal Ideation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Individualized imagery (Experimental)
  Interventions: Behavioral: Individualized imagery
- Control (Active Comparator)
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Individualized imagery — Study personnel will assist participants to create scripts that foster relaxation and safety. Objects, places, and/or scenarios that foster participant relaxation, sense of safety, and/or positive emotions will be identified. Participants will write or type the generated scenario using highly detailed elements (e.g., including visual, olfactory, auditory, tactile, and gustatory sensations, as applicable) associated with the imagery. Study personnel will assist with recording the imagery scripts; audio files will be recorded using an audio recording application. The imagery scripts will be played at night via Bluetooth earbuds connected to the Muse app and script recording while laying down to sleep. The imagery rehearsal prompts will play for approximately 15 minutes, based on 10-20-minute recommendations across imagery rehearsal therapy (IRT) studies
  Arms: Individualized imagery
Behavioral: Control — Participants will wear the earbuds, with use of Muse S headband to collect outcome data without the individualized imagery scripts.
  Arms: Control

SUMMARY:
The purpose of this study is to see how feasible is the use of compact EEG and paired audio technology to administer sleep interventions for inpatients with psychosis, to see if individuals that receive individualized technology-based sleep interventions experience improvements in sleep quality and to see if individuals that receive individualized technology-based sleep interventions experience improvements in symptomatology

ELIGIBILITY:
Inclusion Criteria:

* primary diagnoses of schizophrenia spectrum disorder or mood disorder with psychotic features, as determined by the treatment team or record review
* capacity to consent to the study as determined by licensed psychologists ( or the primary attending psychiatrist
* reported sleep dysfunction which will be determined by a subthreshold or more severe score ≥ 8 on the Insomnia Severity Index (ISI), and/or report experiencing nightmares at least once a week.

Exclusion Criteria:

* primary substance- or medical-induced psychosis
* intellectual and developmental disabilities
* neurodegenerative cognitive disorders
* implanted devices (e.g., Pacemakers)
* on one-to-one supervision or 15-minute safety checks for suicidality or aggression
* patients with roommates that are on 15-minute checks to minimize impact on study participants' awakenings

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-03-05 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility as assessed by coding percentage of use per night (based on duration of physiological measures collected per night divided by hours of sleep) | from start of intervention to end of intervention (upto 80 days after baseline )
Feasibility as assessed by percentage of nights used for the duration of the intervention. | from start of intervention to end of intervention (upto 80 days after baseline )
Feasibility as assessed by a self-report satisfaction survey, Was It Worth It questionnaire | post-intervention(upto 80 days after baseline )
  The measure will consist of 7 items rated on a 5-point Likert scale ranging from Strongly Disagree (1) to Strongly Agree (5), for a maximum score of 35,higher number indicating better satisfaction

SECONDARY OUTCOMES:
Improvements in sleep quality as assessed by the Insomnia Severity Index (ISI) | From Baseline to about 3 months after baseline
  The ISI is an instrument comprising seven questions, and each is scored from 0-7 for a score range of 0-28, a higher number indicating severe clinical insomnia
Improvements in sleep quality as assessed by the Disturbing Dream and Nightmare Severity Index (DDNSI) | From Baseline to about 3 months after baseline
  DDNSI is a 5- item questionnaire. Scoring is done as follows:
  Add nights/per week (0 to 7) + nightmares/week +Q3 which is scored from 0(never/rarely) to 4 (always) +Q4 which is scored from 0 (no problem) to 6 (extremely severe problem) + Q5 which is scored from 0 (not intense) to 6 (extremely severe intensity).Maximum for nightmares/week = 14, so scale is 0 to 14. Score > 10 usually indicate a nightmare disorder.
Improvements in sleep quality as assessed by the Presleep Arousal Scale (PAS) | From Baseline to about 3 months after baseline
  The PAS a 16-item questionnaire and each is scored on a 5-point Likert scale from 1 (not at all) to 5 (extremely), higher number indicating worse outcome
Improvements in sleep quality as assessed by the Dysfunctional Beliefs and Attitudes about Sleep Scale (DBAS) | From Baseline to about 3 months after baseline
  DBAS-16 is a 16-item questionnaire and each question is cored from 0( strongly disagree) to 10 (strongly agree) with higher scores indicating more dysfunctional beliefs and attitudes
Improvements in sleep quality as assessed by the compact electroencephalography (Muse S, Generation 2) | From baseline to end of study (upto 80 days after baseline )
Improvements in symptomology as assessed by the Beck Depression Inventory - II | From Baseline to about 3 months after baseline
  This is a 21-item questionnaire and each is scored from 0-3 for a maximum score of 63, higher score indicating worse outcome
Improvements in symptomology as assessed by the Columbia-Suicide Severity Rating Scale (C-SSRS) | From Baseline to about 3 months after baseline
  Interview administered assessment of suicide ideation and behavior. The interview consists of two subscales, an ideation and behavior subscale. The severity of ideation subscale is rated on a 5-point ordinal scale: 1 = wish to be dead, 2 = nonspecific active suicidal thoughts, 3 = suicidal thoughts with methods, 4 = suicidal intent, and 5 = suicidal intent with plan. The suicidal behavior subscale is rated on a nominal scale that includes actual, aborted, and interrupted attempts; preparatory behavior; and nonsuicidal self-injurious behavior.
Improvements in symptomology as assessed by the abbreviated Positive and Negative Syndrome Scale (PANSS- 6) | From Baseline to about 3 months after baseline
  This is a 6 item questionnaire and each is scored from 1 (Absent) - 7 (Extreme) with a maximum score of 42. The higher the score the greater the symptom severity.
Improvements in symptomology as assessed by the Perceived Stress Questionnaire (PSQ) | From Baseline to about 3 months after baseline
  The PSQ is a 30-item questionnaire and each is scored from e from 1 ("almost never") to 4 ("usually"). Higher scores indicate greater levels of stress
Improvements in symptomology as assessed by the Posttraumatic Checklist for The Diagnostic and Statistical Manual of Mental Disorders (DSM-5) (PCL-5) | From Baseline to about 3 months after baseline
  The PCL-5 is a 20-item questionnaire and each is measured on a 5-point Likert scale from 0(not at all) to 4(extremely), higher number indicating worse outcome

CONTACTS AND LOCATIONS:
Overall Officials: Alia Warner, Ph.D., Principal Investigator — The University of Texas Health Science Center, Houston; Jessica Badawi, Ph.D., Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No